CLINICAL TRIAL: NCT05529277
Title: Dementia Care Management in Der Routineversorgung am Beispiel Der Region Siegen-Wittgenstein (RoutineDeCM)
Brief Title: Implementing Dementia Care Management Into Routine Care in the Region Siegen-Wittgenstein
Acronym: RoutineDeCM
Status: Active, not recruiting | Type: Observational
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Collaborators: University of Siegen (Unknown); Gesundheitsregion Siegerland eG (GRS) (Unknown); Alzheimer Gesellschaft Siegen-Wittgenstein eV (Unknown); Kreisklinikum Siegen (Unknown); Caritasverband Siegen-Wittgenstein eV (Unknown)
Responsible Party: Sponsor
Other Study IDs: GR025; ZMI1-2521FSB907 (Other Grant/Funding Number: Federal Ministery of Health (BMG)); BB110/22 (Other: Ethics Comittee of the Universitymedicine Greifswald)
Record Dates: First submitted 2022-08-26; First posted 2022-09-07 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Dementia; Dementia Alzheimers; Mild Cognitive Impairment; Care Management
MeSH Terms: conditions — Dementia; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dyad of person with cognitive impairment and caregiver: Households identified in routine care receiving a home-based Dementia Care Management.
  Interventions: Other: Dementia Care Management

INTERVENTIONS:
Other: Dementia Care Management — Comprehensive assessment of health care needs of person with cognitive impairment and caregiver followed by algorithm-/ and person-based support in health care planning, implementing and monitoring

SUMMARY:
Dementia Care Management (DeCM) is an evidence-based model of care in Germany. It has proven its efficacy and cost-effectiveness. However it has not been implemented into routine care so far.

The aim of this trial is to implement Dementia Care Management into routine care in a selected region in Germany and evaluate the process of implementation as well as the effect of Dementia Care Management on participants.

Recruited in regular routine care n=60 people with cognitive impairment and/ or their cares will receive Dementia Care Management provided by specifically trained and qualified dementia care managers for 6 months.

Data will be assessed and analysed prior to the implementation, immediately after having received the intervention and at a later time point.

The effect of the intervention on person-oriented health care outcomes wil be analysed as well as factors associated with that.

ELIGIBILITY:
Inclusion Criteria:

* person with cognitive impairment living in household
* living in the region of Siegen-Wittgenstein
* written informed consent

Exclusion Criteria:

* institutionalisation of person with cognitive impairment
* lacking sufficient communication skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People identified in routine care that have a cognitive impairment or live as carerer in a household with a person with cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
unmet needs | 6 months after baseline assessment
  generic standardized assessment implemented as computer-assisted intervention management system (CMS) addresses caregiver burden, medical needs, home care needs, psychosocial needs (depression, sleep quality, pain, hearing, seeing, teeth problems, dementia related problems caused by person with dementia (PwD), medical aids). Adding the needs indicated provides a number of unmet needs.
unmet needs | 12 months after baseline assessment
  generic standardized assessment implemented as computer-assisted intervention management system (CMS) addresses caregiver burden, medical needs, home care needs, psychosocial needs (depression, sleep quality, pain, hearing, seeing, teeth problems, dementia related problems caused by PwD, medical aids). Adding the needs indicated provides a number of unmet needs.

SECONDARY OUTCOMES:
Antidementia drug treatment | 12 months after baseline assessment
  A computer-based home medication review (HMR) encompasses all medications used by the study participants and includes questions about compliance, adverse effects and drug administration. The collection of primary data on medication in the context of the HMR includes both prescription drugs and over-the-counter drugs. The assignment was then integrated using a master file of the Pharmaceutical Index. The following antidementia drugs will be considered: donepezil (N06AD02), rivastigmine (N06AD03), galantamine (N06AD04) and memantine (N06AX01)
Antidementia drug treatment | 6 months after baseline assessment
  A computer-based home medication review (HMR) encompasses all medications used by the study participants and includes questions about compliance, adverse effects and drug administration. The collection of primary data on medication in the context of the HMR includes both prescription drugs and over-the-counter drugs. The assignment was then integrated using a master file of the Pharmaceutical Index. The following antidementia drugs will be considered: donepezil (N06AD02), rivastigmine (N06AD03), galantamine (N06AD04) and memantine (N06AX01)
Neuropsychiatric Symptoms | 6 months after baseline assessment
  Neuropsychiatric Inventory (NPI; Cummings 1997); The NPI represents an interview by proxy on twelve dimensions of neuropsychiatric behaviors, i.e. delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behavior, night-time behavior disturbances, and appetite and eating abnormalities. The presence (0= no, 1= yes) is asked. If present, the severity (rated 1 through 3; mild to severe) and frequency (1 to 4, rarely to very often) of each neuropsychiatric symptom are rated on. Thus the score for each dimension ranges from 0 = not present, 1= mildly and rarely to 12 = severe and often. A total NPI score is calculated as the sum of the frequency by severity scores ofeach domain range: 0 to 144, the higher the more neuropsychiatric symptomatic).
Neuropsychiatric Symptoms | 12 months after baseline assessment
  Neuropsychiatric Inventory (NPI; Cummings 1997); The NPI represents an interview by proxy on twelve dimensions of neuropsychiatric behaviors, i.e. delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behavior, night-time behavior disturbances, and appetite and eating abnormalities. The presence (0= no, 1= yes) is asked. If present, the severity (rated 1 through 3; mild to severe) and frequency (1 to 4, rarely to very often) of each neuropsychiatric symptom are rated on. Thus the score for each dimension ranges from 0 = not present, 1= mildly and rarely to 12 = severe and often. A total NPI score is calculated as the sum of the frequency by severity scores of each domain range: 0 to 144, the higher the more neuropsychiatric symptomatic).
Caregiver Burden | 6 months after baseline assessment
  The revised version of the Zarit-Burden Inventory (ZBI; Zarit et al., 1980) will be used.The revised version ZBI is a caregiver self-report measure to examine burden which is associated with functional/behavioural impairments and home care situation. It contains 22 items using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always).Total scores range from 0 indicating low burden to 88 indicating high burden.
Caregiver Burden | 12 months after baseline assessment
  The revised version of the Zarit-Burden Inventory (ZBI; Zarit et al., 1980) will be used.The revised version ZBI is a caregiver self-report measure to examine burden which is associated with functional/behavioural impairments and home care situation. It contains 22 items using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always).Total scores range from 0 indicating low burden to 88 indicating high burden.

OTHER OUTCOMES:
cognition | 6 months after baseline assessment
  The Mini Mental State Examination (MMSE; Cockrell & Folstein, 1988) will be used. The MMSE is a 30-point questionnaire to measure cognitive impairment. The questions are grouped into seven categories, each representing a different cognitive domain or function: Orientation to time (5 points); Orientation to place (5 points); Registration of three words (3 points); Attention and Calculation (5 points); Recall of three words (3 points); Language (8 points) and Visual Construction (1 point). Scores of 25-30 out of 30 are considered normal; 21-24 as mild, 10-20 as moderate and <10 as severe impairment.
cognition | 12 months after baseline assessment
  The Mini Mental State Examination (MMSE; Cockrell & Folstein, 1988) will be used. The MMSE is a 30-point questionnaire to measure cognitive impairment. The questions are grouped into seven categories, each representing a different cognitive domain or function: Orientation to time (5 points); Orientation to place (5 points); Registration of three words (3 points); Attention and Calculation (5 points); Recall of three words (3 points); Language (8 points) and Visual Construction (1 point). Scores of 25-30 out of 30 are considered normal; 21-24 as mild, 10-20 as moderate and <10 as severe impairment.
frailty | 6 months after baseline assessment
  Frailty will be assessed using the Edmonton frailty scale (EFS; Rolfson et al. 2006) will be used. The EFS is reliable tool in geriatric medicine to assess the frailty of older patients on the domains Cognition, General health status, Functional independence, Social support, Medication use, Nutrition, Mood, Continence and Functional performance.
frailty | 12 months after baseline assessment
  Frailty will be assessed using the Edmonton frailty scale (EFS; Rolfson et al. 2006) will be used. The EFS is reliable tool in geriatric medicine to assess the frailty of older patients on the domains Cognition, General health status, Functional independence, Social support, Medication use, Nutrition, Mood, Continence and Functional performance.
(health-related) quality of life | 6 months after baseline assessment
  Quality of life will be assessed using the the health-related quality of life questionnaire (EQ-5D), a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal.
(health-related) quality of life | 12 months after baseline assessment
  Quality of life will be assessed using EQ-5D, a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal.

CONTACTS AND LOCATIONS:
Overall Officials: Jochen René Thyrian, Prof. Dr., Principal Investigator — German Center for Neurodegenerative Diseases (DZNE); Bernhard Holle, Dr., Principal Investigator — German Center for Neurodegenerative Diseases (DZNE)
Locations (6):
- Germany (6):
  - Deutsches Zentrum für Neurodegenerative Erkrankungen (DZNE), Greifswald, Mecklenburg-Vorpommern
  - University of Siegen, Siegen, North Rhine-Westphalia
  - Caritasverband Siegen-Wittgenstein eV, Siegen, North Rhine-Westphalia
  - Alzheimer Gesellschaft Siegen-Wittgenstein eV, Siegen, North Rhine-Westphalia
  - Kreisklinikum Siegen, Kliniken für Neurologie und Psychiatrie, Siegen, North Rhine-Westphalia
  - Deutsches Zentrum für Neurodegenerative Erkrankungen (DZNE), Witten, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Yes
We will share data upon reasonable request and only aggregated data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: data will become available after end of project - approx. 1/25
Access Criteria: upon reasonable request to the responsible study investigator

REFERENCES:
- [Result] Purwins D, Fahsold A, Quasdorf T, Berthold H, Klas T, Albers B, Seidel K, Haberstroh J, Holle B. Implementation of dementia care management in routine care (RoutineDeCM): a study protocol for process evaluation. BMJ Open. 2023 Aug 23;13(8):e072185. doi: 10.1136/bmjopen-2023-072185. PMID 37612103
- [Result] Seidel K, Rupp L, Thyrian JR, Haberstroh J. Adapting Dementia Care Management to a Regional German Context: Assessment of Changes in Acceptability, Appropriateness, and Feasibility. J Appl Gerontol. 2024 Dec;43(12):1985-1996. doi: 10.1177/07334648241258024. Epub 2024 Jun 5. PMID 38836294
- [Result] Seidel K, Quasdorf T, Haberstroh J, Thyrian JR. Adapting a Dementia Care Management Intervention for Regional Implementation: A Theory-Based Participatory Barrier Analysis. Int J Environ Res Public Health. 2022 Apr 30;19(9):5478. doi: 10.3390/ijerph19095478. PMID 35564877
- [Derived] Thyrian JR, Boekholt M, Boes C, Grond M, Kremer S, Herder-Peyrounette A, Seidel K, Theile-Schurholz A, Haberstroh J. Implementing Dementia Care Management into routine care: protocol for a cohort study in Siegen-Wittgenstein, Germany (RoutineDeCM). BMJ Open. 2024 Jun 26;14(6):e085852. doi: 10.1136/bmjopen-2024-085852. PMID 38926143